CLINICAL TRIAL: NCT00529191
Title: Phase II, Double Blind, Randomized, Placebo-controlled Trial to Evaluate the Safety and Efficacy of Atorvastatin in Subjects With Newly Diagnosed Type 1 Diabetes Mellitus.
Brief Title: Atorvastatin in New Onset Type 1 Diabetes Mellitus (T1DM)
Acronym: TIDM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: FDA Office of Orphan Products Development (U.S. Federal Agency); Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2006-5-4824; R01FD003340 (FDA)
Record Dates: First submitted 2007-09-13; First posted 2007-09-14 (Estimated); Results first posted 2013-03-08 (Estimated); Last update posted 2017-03-13 (Actual); Status verified 2017-01

CONDITIONS: Type 1 Diabetes
Keywords: Type I Diabetes (T1DM); Atorvastatin (Lipitor); Insulin; Pancreas; Beta Cells
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Insulin Resistance | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Atorvastatin (Experimental): Two out of every three patients will receive atorvastatin.
  Interventions: Drug: Atorvastatin
- Placebo (Placebo Comparator): One out of three subjects will receive a placebo.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Atorvastatin — Pill, initially at 10 mg, then after 4 weeks, 20 mg Once daily for a total of 12 months
  Other Names: Lipitor
  Arms: Atorvastatin
Other: Placebo — One out of three subjects will receive a placebo.
  Arms: Placebo

SUMMARY:
The goal of this application is to evaluate the safety and efficacy of atorvastatin as a potential treatment to preserve beta cell function in children and young adults with newly diagnosed type 1 diabetes (T1DM).

DETAILED DESCRIPTION:
Type 1 diabetes is an autoimmune disease that is characterized by destruction of the insulin-producing beta cells of the pancreas. T1DM therapy requires insulin administration, either by multiple daily injections or by insulin pump. However, in many patients, blood sugar control remains suboptimal and complications develop that shorten life expectancy and severely impact quality of life. At the time of diagnosis, most patients still have significant residual beta cell function. Previous research has shown that weakening the immune system's attack on the pancreatic beta cells may help to preserve or potentially increase insulin production.

Preliminary studies have shown that members of the statin family of medications, including atorvastatin (Lipitor®), preserve beta cell function in a mouse model of type 1 diabetes. These finding suggest that use of atorvastatin in combination with insulin therapy may delay and potentially reverse the destruction of beta cells in patients who have recently developed type 1 diabetes. Atorvastatin (Lipitor®) is approved for use in adults and children (>10 years of age) who have elevated blood cholesterol levels. This study will examine whether atorvastatin (Lipitor®) may also help the body preserve insulin production in patients with newly diagnosed (within 8 weeks) type 1 diabetes.

Patients will be randomly assigned to take either atorvastatin (Lipitor®) or placebo. Two out of every 3 patients will receive atorvastatin and 1 out of 3 will get placebo. As this is a double-blinded study, neither the care team nor the patient will know if they are actually taking atorvastatin (Lipitor®). Patients who have given consent to participate in the study and pass the required screening tests will take the assigned treatment every day for 12 months. All patients will begin taking 10 mg once daily, the recommended starting dose. After 4 weeks, the dose will be increased to 20 mg. In addition to a high standard of diabetes care and the medication, patients will have blood tests during 7 visits over an 18 month period.

ELIGIBILITY:
Inclusion Criteria:

* Individuals 10-19 years of age (Tanner Stage II or greater),
* The presence of one or more serum antibodies to islet cell proteins (anti- glutamic acid decarboxylase [GAD], islet antigen 2 or insulin autoantibodies) as assessed in standard practice,
* Diagnosis of T1DM within the 8 weeks prior to study entry
* Peak stimulated C-peptide level >0.2pmol/mL following mixed meal tolerance test (MMTT) performed at least 3 weeks after diagnosis,
* Females of reproductive potential must not plan on conceiving a child during the treatment program, and agree to use a medically accepted form of contraception

Exclusion Criteria:

* Subjects currently receiving cyclosporine, fibric acid derivatives, niacin (nicotinic acid), erythromycin, clarythromycin, nefazodone, itraconazole, ketoconazole or protease inhibitors,
* Pregnancy or breast-feeding,
* Clinical AIDS, AIDS related syndrome (ARS) or known positive HIV serology,
* Subjects treated with immunosuppressive therapy in the past 12 months,
* Subjects receiving glucocorticoid therapy or therapy other than insulin that is likely to affect glucose homeostasis (such as sulfonylureas, thiazolidinediones, metformin or amylin),
* Subjects with other autoimmune diseases, except autoimmune thyroid disease,
* Subjects with any illness that might complicate diabetes management or preclude treatment with atorvastatin,
* Transplant recipients,
* Evidence of liver dysfunction or myopathy

Ages: 10 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2007-07; Primary Completion 2011-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven M Willi, M.D, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Diabetes Center for Children & Clinical Translational Research Center, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share these data, except in aggregate.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from medical clinics at CHOP from July 2007- January 2010
Groups:
- Atorvastatin: Two out of every 3 patients will receive atorvastatin in tablet form. The subject will start on 10mg of atorvastatin daily for four weeks, and then titrate up to 20mg daily. There will be 12 months of treatment followed by 6 months of a washout period.
- Placebo: Placebo treated. Patients will receive tablets daily.There will be 12 months of treatment followed by 6 months of a washout period.
Period: Overall Study
Arm/Group | Atorvastatin | Placebo
Started | 27 | 13
Completed | 24 | 13
Not Completed | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Atorvastatin: Two out of every 3 patients will receive atorvastatin.
- Placebo: Placebo treatment
- Total: Total of all reporting groups
Arm/Group | Atorvastatin | Placebo | Total
Number analyzed (Participants) | 27 | 13 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 26 | 12 | 38
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.38 (1.96) | 13.30 (2.03) | 13.33 (2.055)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 9 | 20
  Male | 16 | 4 | 20
Region of Enrollment [Number; unit: participants]
  United States | 27 | 13 | 40

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of a Daily Dose of Atorvastatin to Maintain Islet Cell Function as Measured by a 4-hour C-peptide Area Under Curve (AUC) in Patients With Newly Diagnosed Type 1 Diabetes Mellitus
Description: The change in C-peptide measurements collected over a 4 hour period (0, 30, 60, 90, 120, 150, 180, 210 and 240 minutes) after a Mixed Meal Tolerance Test at baseline vs 12 months post-treatment were calculated. The area under the curve for these combined measurements is calculated and the unit of measure is nanogram x minutes / mL. Efficacy (success) is defined by < 7.5% reduction in AUC for 4-hr MMTT.
Time Frame: Baseline vs 12-month
Population: Participants who completed their 12-month treatment were included in the analysis, in which the change in C-peptide AUC at baseline and 12-months were calculated. Efficacy (success) is defined by < 7.5% reduction in AUC for 4-hr MMTT.
Measure: Mean (Standard Deviation); unit: nanogram*minutes/ml
Arm/Group | Atorvastatin | Placebo
Number analyzed (Participants) | 27 | 13
nanogram*minutes/ml | 345 (679) | 178 (308)

2. Secondary Outcome: % Subjects Without Change in 2-hour C-peptide AUC in Response to the MMTT at Baseline vs. 12 Months
Description: The C-peptide AUC measurements are collected over a 2 hour period (with 30 minute intervals) after a Mixed Meal Tolerance Test. The area under the curve from these combined measurements (from 0 to 120 or 0 to 240 minutes) is calculated and the unit of measure is nanogram*minutes/ml. The change in C-peptide AUC in response to a 2 hour MMTT at baseline vs 12 months were calculated, and efficacy (success) is defined as < 7.5% reduction.
Time Frame: Baseline vs 12 months
Measure: Number; unit: % of participants with efficacy
Arm/Group | Atorvastatin | Placebo
Number analyzed (Participants) | 27 | 13
% of participants with efficacy | 14.8 | 38.4

3. Secondary Outcome: Mean Daily Insulin Dose Per kg Body Weight for 7 Days
Description: Mean daily insulin dose per kg body weight for the 1 week preceding each scheduled study visit.
Time Frame: Visit 1, 2, 3, 4, 5, 6, 7
Measure: Mean (Standard Deviation); unit: units/kg
Arm/Group | Atorvastatin | Placebo
Number analyzed (Participants) | 27 | 13
units/kg
  Visit 1 | 0.53 (0.26) | 0.62 (0.26)
  Visit 2 | 0.50 (0.25) | 0.52 (0.22)
  Visit 3 | 0.48 (0.21) | 0.50 (0.26)
  Visit 4 | 0.59 (0.21) | 0.47 (0.30)
  Visit 5 | 0.64 (0.22) | 0.59 (0.35)
  Visit 6 | 0.65 (0.24) | 0.64 (0.36)
  Visit 7 | 0.70 (0.35) | 0.71 (0.34)

4. Secondary Outcome: Levels of HbA1c at Months 3, 6, 9, 12 and 18
Time Frame: 3, 6, 9, 12, and 18 months
Measure: Mean (Standard Deviation); unit: percentage of glycated hemoglobin
Arm/Group | Atorvastatin | Placebo
Number analyzed (Participants) | 27 | 13
percentage of glycated hemoglobin
  3 months | 6.68 (0.95) | 6.39 (0.95)
  6 months | 7.13 (0.90) | 6.62 (1.22)
  9 months | 7.47 (1.44) | 6.86 (0.91)
  12 months | 7.38 (1.19) | 7.26 (1.45)
  18 months | 8.04 (1.82) | 7.94 (2.62)

5. Secondary Outcome: Blood Glucose Control (Number of Participants With Hypoglycemia)
Description: Blood glucose control as determined from home glucose meter downloads for the 1 week preceding the visit. The number of subjects with hypoglycemic episodes requiring treatment (BG < 70 mg/dl)
Time Frame: Baseline, Month 12, Month 18
Population: All participants contributing data
Measure: Count of Participants; unit: Participants
Groups:
- Atorvastatin: Participants in Atorvastatin arm who had hypoglycemic episodes requiring treatment
  Two out of every three patients will receive atorvastatin.
  Atorvastatin: Pill, initially at 10 mg, then after 4 weeks, 20 mg Once daily for a total of 12 months
- Placebo: Participants in placebo arm who had hypoglycemic episodes requiring treatment
  Placebo treated. Patients will receive tablets daily.There will be 12 months of treatment followed by 6 months of a washout period.
Arm/Group | Atorvastatin | Placebo
Number analyzed (Participants) | 27 | 13
Participants
  Baseline | 16 | 7
  12 Month | 16 | 9
  18 Month | 8 | 8

6. Secondary Outcome: Number of Episodes of Hypoglycemia Requiring Any Treatment
Description: number of episodes of hypoglycemia requiring any treatment, defined by the need for treatment with glucagon or third party intervention.
Time Frame: Baseline, Month 12, Month 18
Population: All subjects contributing data
Measure: Mean (Standard Deviation); unit: episodes
Arm/Group | Atorvastatin | Placebo
Number analyzed (Participants) | 27 | 13
episodes
  Baseline: number analyzed (Participants) | 16 | 7
  Baseline | 4.13 (3.95) | 2.86 (3.98)
  Month 12: number analyzed (Participants) | 16 | 9
  Month 12 | 3.44 (3.01) | 2.44 (2.51)
  Month 18: number analyzed (Participants) | 8 | 8
  Month 18 | 2.75 (3.65) | 2.5 (2.2)

7. Secondary Outcome: Study Drug Compliance Rate Overall
Description: Compliance is defined as >=80% expected dosage consumed during the visit period.
Time Frame: 12 months treatment
Measure: Number; unit: % of compliant participants
Arm/Group | Atorvastatin | Placebo
Number analyzed (Participants) | 27 | 13
% of compliant participants | 85.1 | 76.9

8. Secondary Outcome: HDL and LDL Cholesterol Levels in Participants Stratified by the Preservation of Islet Cell Function
Description: Relationship between atorvastatin's effect on HDL and LDL cholesterol and the preservation of islet cell function.
  Islet cell preservation defined as: <7.5% Reduction in C-Pep
Time Frame: Baseline, Week 1, Month 3, Month 6, Month 9, Month 12,
Measure: Mean (Standard Deviation); unit: mg/dl
Groups:
- Atorvastatin NO Islet Cell Preservation; Atorvastatin YES Islet Cell Preservation: Two out of every three patients will receive atorvastatin.
  Atorvastatin: Pill, initially at 10 mg, then after 4 weeks, 20 mg Once daily for a total of 12 months
- Placebo NO Islet Cell Preservation; Placebo YES Islet Cell Preservation: Placebo treated. Patients will receive tablets daily.There will be 12 months of treatment followed by 6 months of a washout period.
Arm/Group | Atorvastatin NO Islet Cell Preservation | Placebo NO Islet Cell Preservation | Atorvastatin YES Islet Cell Preservation | Placebo YES Islet Cell Preservation
Number analyzed (Participants) | 24 | 8 | 3 | 5
mg/dl
  Baseline- HDL Cholesterol (mg/dL) | 47.58 (16.39) | 44.75 (18) | 47.33 (2.31) | 53.2 (16.39)
  Baseline - LDL Cholesterol (mg/dL) | 99.04 (22.37) | 96.13 (22.99) | 83.67 (25.97) | 99 (13.04)
  Week 1- HDL Cholesterol (mg/dL) | 45.43 (14.33) | 48.25 (14.26) | 52.33 (5.69) | 47.2 (13.88)
  Week 1 - LDL Cholesterol (mg/dL) | 68.91 (16.4) | 97.63 (17.9) | 57.67 (12.06) | 86.4 (12.46)
  Month 3- HDL Cholesterol (mg/dL) | 45.05 (14.49) | 48.25 (18.69) | 43.33 (4.04) | 49.25 (12.31)
  Month 3 - LDL Cholesterol (mg/dL) | 61 (20.88) | 106.25 (18.44) | 48 (12.17) | 91.5 (20.21)
  Month 6- HDL Cholesterol (mg/dL) | 48 (16.07) | 50.5 (20.7) | 51.67 (5.51) | 54.75 (19.47)
  Month 6 - LDL Cholesterol (mg/dL) | 63.1 (24.52) | 102.5 (16.21) | 54 (7) | 96.75 (20.93)
  Month 9- HDL Cholesterol (mg/dL) | 49.1 (14.86) | 45.88 (12.57) | 55.33 (11.15) | 50 (21.71)
  Month 9 - LDL Cholesterol (mg/dL) | 67.24 (24.7) | 97 (4.17) | 65.33 (28.01) | 90.75 (8.06)
  Month 12 - HDL Cholesterol (mg/dL) | 47.95 (14.49) | 45.75 (16.34) | 57.33 (14.15) | 47 (8.31)
  Month 12 - LDL Cholesterol (mg/dL) | 61.52 (20.04) | 102.75 (20.9) | 66 (23.64) | 96.4 (6.66)

ADVERSE EVENTS:
Time Frame: Events were reported over the one year treatment phase of the study.
Description: Adverse events were reported or observed at interim visits, and were systematically collected.
Arm/Group | Atorvastatin | Placebo
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/13
Other Adverse Events (participants affected / at risk) | 23/27 | 10/13
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atorvastatin (N=27) | Placebo (N=13)
Hypoglycemia (Endocrine disorders) | 3 (3) | 0 (0)
Headache (Nervous system disorders) | 7 (11) | 3 (3) — Patient report of headache at interim assessment.
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (4) — Reported or observed at interim visit.
Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 9 (11) | 4 (7) — Respiratory Infection reported or observed at interim visit.
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (2) — Reported or observed at interim visit.
Nausea (Gastrointestinal disorders) | 4 (5) | 2 (2) — Reported or observed at interim visit.
Fever (General disorders) | 8 (11) | 2 (2) — Reported or observed at interim visit.
Gastroenteritis (Gastrointestinal disorders) | 4 (4) | 2 (2) — Reported or observed at interim visit.
Diarrhea (Gastrointestinal disorders) | 1 (1) | 2 (2) — Reported or observed at interim visit.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No